CLINICAL TRIAL: NCT03338387
Title: Acipimox Administration Together With Short-Term Exercise Exerts A Co-Feedback of Growth Hormone, Pancreatic Polypeptide, Peptide YY and Leptin on Ghrelin in Young Bulimic Czech Women: A Randomized Study
Brief Title: Co-Feedback Action of Growth Hormone, PP and PYY on Ghrelin in Bulimia
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kvido Smitka, M.D., Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZV Grant Agency
Record Dates: First submitted 2017-10-06; First posted 2017-11-09 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Eating Disorder; Bulimia Nervosa
Keywords: neuropeptides; microdialysis
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa | interventions — acipimox

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acipimox (Experimental): Other Names: Olbetam
  Interventions: Drug: Acipimox
- Placebo (Placebo Comparator): Other Names:
  Placebo (for Olbetam)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acipimox — Acipimox
  Other Names: 5-methylpyrazine-2-carboxylic acid 4-oxide
  Arms: Acipimox
Drug: Placebo — Placebo Other Names: Placebo (for Olbetam)
  Other Names: Cellulose pills manufactured to mimic Acipimox 250Mg Capsule
  Arms: Placebo

SUMMARY:
This study evaluates the addition of Acipimox or placebo to exercise on growth hormone release and ghrelin secretion in bulimic patients and in healthy women. Two groups of participants will receive Acipimox together with exercise versus identical placebo with exercise.

DETAILED DESCRIPTION:
Acipimox and exercise each increase growth hormone release, but they do so by different mechanisms.

Acipimox is an anti-lipolytic drug and increases growth hormone release by decreasing free fatty acids levels and that Acipimox may exert to a negative feedback of growth hormone on ghrelin.

Physical exercise is a potent physiological stimulus for growth hormone release. As ghrelin has a stimulatory effect on growth hormone secretion, growth hormone may inhibit circulating ghrelin levels via a feedback loop. Growth hormone stimulates lipolysis and resultant free fatty acids may suppress ghrelin secretion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of bulimia nervosa
* Body mass index (BMI) between 18 and 23 kg/m2

Exclusion Criteria:

* History of heart disease
* History of bleeding disorders
* Subjects with diabetes type 1 or 2, hypo- or hyperthyroidism
* Subjects with hepatogastroenteric disease
* Pregnant, trying to become pregnant or breast feeding
* Patients with other psychiatric diseases

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2003-05-06 (Actual); Primary Completion 2007-12-16 (Actual); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma growth hormone levels | baseline and over a total 2 weeks
  Plasma growth hormone (mIU/L) levels will be measured by a commercial RIA kit in the morning and after exercise alone or together with Acipimox administration over a total of 2 weeks.

SECONDARY OUTCOMES:
Changes in extracellular adipose tissue glycerol levels | baseline and over a total 2 weeks
  Extracellular adipose tissue glycerol (umol/L) levels will be measured using microdialysis technique and analyzed with a radiometric kit in the morning and after exercise alone or together with Acipimox administration over a total of 2 weeks.

OTHER OUTCOMES:
Changes in body mass index (BMI) | baseline and over a total 2 weeks
  Weight in kilograms and height in meters will be measured in the morning and after exercise alone or together with Acipimox administration over a total of 2 weeks. Weight and height will be combined to report BMI in kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Kvido Smitka, M.D., Ph.D., Principal Investigator — Charles University, Czech Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nedvidkova J, Smitka K, Papezova H, Vondra K, Hill M, Hainer V. Acipimox during exercise points to an inhibitory feedback of GH on ghrelin secretion in bulimic and healthy women. Regul Pept. 2011 Feb 25;167(1):134-9. doi: 10.1016/j.regpep.2010.12.012. Epub 2011 Jan 13. PMID 21237212
- [Background] Smitka K, Papezova H, Vondra K, Hill M, Hainer V, Nedvidkova J. A higher response of plasma neuropeptide Y, growth hormone, leptin levels and extracellular glycerol levels in subcutaneous abdominal adipose tissue to Acipimox during exercise in patients with bulimia nervosa: single-blind, randomized, microdialysis study. Nutr Metab (Lond). 2011 Nov 17;8(1):81. doi: 10.1186/1743-7075-8-81. PMID 22093818
- [Background] Smitka K, Papezova H, Vondra K, Hill M, Hainer V, Nedvidkova J. Short-term exercise combined with Acipimox administration induces an increase in plasma ACTH and its subsequent fall in the recovery phase in bulimic women. Regul Pept. 2013 Mar 10;182:45-52. doi: 10.1016/j.regpep.2012.12.010. Epub 2013 Jan 11. PMID 23318497
- [Background] Smitka K, Papezova H, Vondra K, Hill M, Hainer V, Nedvidkova J. The role of "mixed" orexigenic and anorexigenic signals and autoantibodies reacting with appetite-regulating neuropeptides and peptides of the adipose tissue-gut-brain axis: relevance to food intake and nutritional status in patients with anorexia nervosa and bulimia nervosa. Int J Endocrinol. 2013;2013:483145. doi: 10.1155/2013/483145. Epub 2013 Sep 9. PMID 24106499
- [Background] Smitka K, Maresova D. Adipose Tissue as an Endocrine Organ: An Update on Pro-inflammatory and Anti-inflammatory Microenvironment. Prague Med Rep. 2015;116(2):87-111. doi: 10.14712/23362936.2015.49. PMID 26093665
- [Background] Smitka K, Nedvidkova J, Vondra K, Hill M, Papezova H, Hainer V. Acipimox Administration With Exercise Induces a Co-feedback Action of the GH, PP, and PYY on Ghrelin Associated With a Reduction of Peripheral Lipolysis in Bulimic and Healthy-Weight Czech Women: A Randomized Study. Front Endocrinol (Lausanne). 2019 Mar 12;10:108. doi: 10.3389/fendo.2019.00108. eCollection 2019. PMID 30915029
- [Background] Roubalova R, Prochazkova P, Papezova H, Smitka K, Bilej M, Tlaskalova-Hogenova H. Anorexia nervosa: Gut microbiota-immune-brain interactions. Clin Nutr. 2020 Mar;39(3):676-684. doi: 10.1016/j.clnu.2019.03.023. Epub 2019 Mar 23. PMID 30952533
- [Background] Smitka K, Prochazkova P, Roubalova R, Dvorak J, Papezova H, Hill M, Pokorny J, Kittnar O, Bilej M, Tlaskalova-Hogenova H. Current Aspects of the Role of Autoantibodies Directed Against Appetite-Regulating Hormones and the Gut Microbiome in Eating Disorders. Front Endocrinol (Lausanne). 2021 Apr 19;12:613983. doi: 10.3389/fendo.2021.613983. eCollection 2021. PMID 33953692
- [Background] Prochazkova P, Roubalova R, Dvorak J, Kreisinger J, Hill M, Tlaskalova-Hogenova H, Tomasova P, Pelantova H, Cermakova M, Kuzma M, Bulant J, Bilej M, Smitka K, Lambertova A, Holanova P, Papezova H. The intestinal microbiota and metabolites in patients with anorexia nervosa. Gut Microbes. 2021 Jan-Dec;13(1):1-25. doi: 10.1080/19490976.2021.1902771. PMID 33779487